CLINICAL TRIAL: NCT00537199
Title: Evaluation of OraTest in Combination With Visual Examination in the Improved Detection of Oral Mucosal Lesions Suspicious of Serious Pathology in High-Risk Patients for the Purpose of Referral to the Health Care Professional Experienced in Oral Cancer: Phase III Clinical Trial Comparing the Sensitivity and Assessing the Specificity of OraTest in Combination With Visual Examination and Visual Examination Alone in Patients at High Risk as Defined by Age and Lifestyle Factors (ZIL-401)
Brief Title: OraTest in Combination With Visual Examination and Visual Examination Alone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early as per request by sponsor, Zila Biotechnology, Inc.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Zila Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-1008
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2009-12

CONDITIONS: Head And Neck Cancer; Oropharynx Cancer
Keywords: Head And Neck; Oropharynx; Oral Cancer; OraTest; OraTest Dye; Rinse Staining Procedure; Visual Examination
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OraTest + Visual Exam (Other): OraTest dye
  Interventions: Other: Visual Examination; Drug: OraTest

INTERVENTIONS:
Other: Visual Examination — Two (2) scheduled visits for visual examination of mouth for abnormal lesions and glands in the neck.
Drug: OraTest — Two (2) scheduled visits for rinse staining: 2 teaspoons of OraTest for 20 seconds, then spit.
  Other Names: OraTest Dye; Rinse Staining Procedure

SUMMARY:
Primary Objectives:

1. To assess the ratio in sensitivities of OraTest® in combination with visual examination versus visual examination alone in the detection of serious pathology defined as severe dysplasia, CIS, or cancer of the O/OP cavity in patients who are at high risk for squamous cell carcinoma, carcinoma in situ, or severe dysplasia of the oral/oropharyngeal (O/OP) cavity due to their age and lifestyle risk factors.
2. To estimate the adjusted specificity of OraTest® in combination with visual examination in the detection of severe dysplasia, CIS, or cancer of the O/OP cavity.

Secondary Objectives:

1. To assess the ratio of sensitivity of OraTest® in combination with visual examination versus visual examination alone in the detection of certain chromosomal abnormalities (17p chromosomal deletions, or both 3p and 9p chromosomal deletions), severe dysplasia, CIS, or cancer of the O/OP cavity in patients who are at high risk for squamous cell carcinoma, carcinoma in situ, or severe dysplasia of the oral/oropharyngeal (O/OP) cavity due to their age and lifestyle risk factors.
2. To obtain the adjusted specificity of OraTest® in combination with visual examination in the detection of certain chromosomal abnormalities (17p chromosomal deletions, or both 3p and 9p chromosomal deletions), severe dysplasia, CIS or cancer of the O/OP cavity.
3. To evaluate the chromosomal status of the positively staining lesions with respect to 3p, 9p, or 17p deletions.
4. To carry out gene expression studies on biopsies and map these onto an analysis of the widespread chromosomal imbalances in stain-positive and stain-negative lesions.
5. To evaluate the quantitative and qualitative toxicities, as well as other safety parameters, of tolonium chloride 5 mg/mL (OraTest®).

DETAILED DESCRIPTION:
OraTest® is a blue dye that is designed to stain cancer cells differently than normal cells.

SCHEDULED EVALUATION (FIRST VISIT):

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your medical history will be recorded. Women who are able to have children must have a negative urine pregnancy test. Your heart rate, breathing, temperature, and blood pressure will be measured before as well as after the first visit.

Visual Exam - If you are found to be eligible to take part in this study, you will have a visual examination where a doctor (Examiner #1) will look inside your mouth very carefully to look for any abnormal lesions and check the glands in your neck. This is called the visual exam.

Rinse Staining Procedure (OraTest®) - A second doctor (Examiner #2) will perform another oral exam, followed by the new test using OraTest®. This new test uses a blue dye which may stain any potential cancer blue so it may make it easier for the doctor to detect any abnormal lesions in your mouth. You will be asked not to have intensely-colored sweets like lollipops or drinks like black currant juice within 24 hours of your scheduled visit. First you will rinse your mouth with about 6 teaspoons of vinegar solution for about 20 seconds and spit it out. Next you will rinse your mouth with 6 teaspoons of water for 20 seconds and spit it out. Then you will rinse your mouth with about 2 teaspoons of OraTest® for 20 seconds and spit it out. Then you will rinse your mouth with about 6 teaspoons of vinegar solution for 20 seconds and then spit it out. Then you will rinse your mouth with 6 teaspoons of water for 20 seconds and spit it out. Examiner 2 will then check and see if any abnormal tissue absorbed the dye.

If no suspicious lesions are found by either doctor, you will have completed the study. You will be asked to notify the clinic, by phone, if any side effects occur within 7 days after your visit. If you are unable to phone the clinic, you will be given diary cards to record these side effects. The diary cards are to be mailed to the doctor in the pre-stamped envelope given to you.

If any suspicious lesions are found by either doctor (or both), then you will be asked to return in about 2 weeks to confirm the result. This is called the Confirmation Exam.

CONFIRMATION EXAM (SECOND VISIT):

At the visit to confirm the result, you will be examined by the same doctor(s) who found the suspicious lesion(s). The doctor(s) will use the same examination method that was used during the first visit. Your heart rate, breathing, temperature, and blood pressure will be measured before as well as after the second visit.

If you have any suspicious lesions, a specialist at M. D. Anderson will biopsy your lesion(s), at this second visit or within 5 days after the visit. During the biopsy, the doctor may use the OraTest® cotton swab to help locate the suspicious spot. If the dye is used at the biopsy visit, your heart rate, breathing, temperature, and blood pressure will be measured before and after the use of OraTest®. After locating the spot, the doctor will perform the biopsy. This means that some tissue lining in your mouth from the suspicious area will be removed. Some of your tissue will be sent to a laboratory for diagnosis. Your doctor will decide the type of care you may need based on the results of the biopsy. The biopsy procedure is standard practice and may happen even if you did not participate in this study. After the biopsy is taken of the lesion, you will have completed the study.

If a suspicious lesion is found and you are required to have a biopsy, a sample of tissue from the biopsy will be sent to a laboratory outside of M.D. Anderson for review and diagnosis. Medical research including genetic testing, chromosomal analysis and other tests may be performed on your biopsy. These samples cannot be returned to you because the tissue is destroyed during the genetic tests. Before your tissue is sent to the outside laboratory your name and any personal identifying information will be coded to protect your privacy. M. D. Anderson will not have oversight of any leftover tissue and/or blood that will be banked by BRT Laboratories Inc. for additional research.

If no suspicious lesions are seen at this second visit, then you have completed the study. If the dye was used during the exam, then you will be asked to notify the clinic by phone if any side effects occur within 7 days after your visit. If you are unable to phone the clinic, you will be given diary cards to record these side effects. The diary cards are to be mailed to the doctor in the pre-stamped envelope given to you.

This is an investigational study. OraTest® has not yet been FDA approved for commercial use. All study procedures and OraTest® will be provided free of charge; the Sponsor will pay for the study drug and pregnancy test if necessary. If further standard of care is needed (for example, due to abnormalities found), you and/or your insurance company will be responsible for the cost. Insurance companies and Medicare may not pay for the costs of some research studies like this one. If your insurance company does not cover the cost of care, then you will have to pay these costs. You have the right to ask what it will cost you to take part in this study or to have other treatments. If you withdraw from the study early, you will only be paid for the portion of the study that you completed. Up to 4000 patients will take part in this multicenter study. Up to 50 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. High risk of oral cancer as defined by a twenty-pack/year cigarette smoking history or equivalent and is either a current smoker or has quit smoking within the last 24 months. Twenty-pack/year equivalent is defined as ½ pack/day for 40 years, or one pack/day for 20 years, or 2 packs/day for 10 years, or 4 packs/day for 5 years. AND/OR;
2. Ten-year history of twenty orally-consumed alcohol units/week and is either a current drinker or has quit drinking within the last 24 months. Twenty orally-consumed alcohol units/week is defined as the equivalent of twenty - 1 ounce shots of whisky or spirits/week (20 ounces = 600 mL), or twenty - 3 ounce glasses of wine/week (60 ounces = 1800 mL), or twenty - 12 ounce glasses of beer/week (240 ounces = 7200 mL);
3. Male or female, at least 45 years of age;
4. Written informed consent.
5. Females of childbearing potential may be enrolled following a negative urine pregnancy test performed at the SE visit. Abstinence will be considered an acceptable form of birth control.

Exclusion Criteria:

1. History of oral cancer, surgery or biopsy for suspected oral neoplasm;
2. History of recent oral surgery, periodontal treatment, or oral trauma (<14 days) or current orthodonture (e.g., braces);
3. Known hypersensitivity to study drug or its analogs;
4. Active and uncontrolled infection or any other severe concurrent disease that in the judgment of the investigator would make the patient inappropriate for entry into this study;
5. Psychiatric disorders which would interfere with informed consent or follow-up;
6. Use of any investigational agent within previous 30 days;
7. Female that is lactating or demonstrating positive pregnancy test;
8. Patients in whom betel nut use/abuse has been reported within the past 5 years;
9. Patients currently taking medication containing prohibited dyes.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chambers, DMD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/04/07 through 06/22/07. Single participant recruited at UT MD Anderson Cancer Center although multi-center study.
Pre-assignment Details: Only 1 patient enrolled prior to sponsor Zila Biotechnology terminating study. Study monitoring done by sponsor; no final data available on part of University of Texas (UT) MD Anderson Cancer Center.
Groups:
- OraTest + Visual Exam: Visual oral exam, followed by OraTest Rinse Staining Procedure
Period: Overall Study
Arm/Group | OraTest + Visual Exam
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | OraTest + Visual Exam
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 64 [64 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratio (Percentage) of Sensitivity of OraTest + Visual Exam Versus Sensitivity of Visual Exam Alone
Description: Primary efficacy parameters, ratio of sensitivity of OraTest® in combination with visual exam versus visual exam alone is the difference between the adjusted specificity for OraTest in combination with visual exam and the adjusted specificity for visual exam alone.
  Reported ratio as percentage of patients with abnormalities (suspicious lesions) found upon visual exam of the mouth with and without OraTest® dye.
Time Frame: Following two (2) scheduled visits for visual examination, up to one month following first exam
Population: No analysis was performed. Study was terminated by sponsor.
Arm/Group | OraTest + Visual Exam
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection from first exam to confirmation exam two weeks later, followed up to one month.
Description: Study was terminated after first patient enrolled.
Arm/Group | OraTest + Visual Exam
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination by sponsor resulted in only 1 patient enrolled and no analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No